CLINICAL TRIAL: NCT06262516
Title: Randomized-Controlled Trial Examining Oncologic and Perioperative Outcomes for Nephroureterectomy With and Without Lymph Node Dissection for Upper Tract Urothelial Cell Carcinoma
Brief Title: Nephroureterectomy With and Without Lymph Node Dissection for Upper Tract Urothelial Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE2824
Record Dates: First submitted 2024-02-06; First posted 2024-02-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Urothelial Carcinoma
Keywords: Nephroureterectomy; Kidney and ureter; Upper Tract Urothelial Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Nephroureterectomy; Lymph Node Excision

STUDY DESIGN:
Intervention Model Description: This study is designed as a 1:1 two armed randomized-controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nephroureterectomy With Lymph Node Dissection (Experimental): Participants will undergo nephroureterectomy for UTUC and will receive LND.
  Interventions: Procedure: Nephroureterectomy; Procedure: Lymph Node Dissection
- Nephroureterectomy Without Lymph Node Dissection (Active Comparator): Participants will undergo nephroureterectomy for UTUC and will not receive LND.
  Interventions: Procedure: Nephroureterectomy

INTERVENTIONS:
Procedure: Nephroureterectomy — Participants will undergo standard-of-care nephroureterectomy for UTUC.
Procedure: Lymph Node Dissection — Participants will receive lymph node dissection alongside nephroureterectomy for UTUC.
  Arms: Nephroureterectomy With Lymph Node Dissection

SUMMARY:
The goal of this study is to conduct the first randomized-controlled trial to determine the oncologic efficacy of lymph node dissection in participants with upper tract urothelial cell carcinoma. The main questions it aims to answer are:

* To determine oncologic outcomes, specifically 2-year recurrence-free survival
* To determine other oncologic outcomes including treatment-free, cancer-specific and overall survival
* To determine time to recurrence and recurrence patterns
* To determine use of adjuvant therapies
* To determine perioperative complications

Participants will undergo nephroureterectomy with or without lymph node dissection. Researchers will compare these two groups to determine the oncologic efficacy of performing lymph node dissection.

DETAILED DESCRIPTION:
Upper Tract Urothelial Carcinoma (UTUC) is a rare disease with complex management. Some participants with clinically negative nodes may still receive a lymph node dissection (LND) with nephroureterectomy, and currently, no randomized controlled trial exists to evaluate the oncologic efficacy of this practice. According to current American Urologic Association guidelines, Nephroureterectomy is the standard of care intervention for high-risk UTUC and low-risk UTUC is endoscopically unresectable. The aim of the present study is to determine the efficacy, specifically 2-year recurrence-free survival, of lymph node dissection at time of nephroureterectomy for participants with UTUC, compared to no lymph node dissection, as well as examine other oncologic outcomes and complication rates

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Diagnosis of UTUC as determined by upper tract biopsy (either low or high grade)
* Planned for nephroureterectomy by their urologic surgeon
* Disease that is ≤cT4, N0M0. Participants must have complete TNM staging prior to surgery. cT disease can be determined by biopsy of the mass (if biopsy was deep enough) or imaging (CT/MRI). cN and cM stage must be determined by preoperative imaging of the chest, abdomen and pelvis.
* No concomitant muscle-invasive bladder cancer
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pathologically enlarged lymph nodes suspicious for metastases which would require lymph node dissection regardless of trial (>cN0)
* Presence of distant metastases
* Concomitant muscle invasive bladder cancer
* The participant is in a reduced general condition or has a life-threatening disease.
* The participant has a psychiatric disorder that precludes them from understanding the consent process.
* The patient is pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 2 years post-op
  Kaplan-Meier will compare recurrence-free survival time between participants who received LND vs participants who did not receive LND.

SECONDARY OUTCOMES:
Treatment-free survival | 2 years post-op
  Kaplan-Meier will compare treatment-free survival time between participants who received LND vs participants who did not receive LND.
Cancer-specific survival | 2 years post-op
  Kaplan-Meier will compare cancer-specific survival time between participants who received LND vs participants who did not receive LND.
Overall Survival | 2 years post-op
  Kaplan-Meier will compare the overall survival between participants who received LND vs participants who did not receive LND.
Time to recurrence | 2 years post-op
  Kaplan-Meier will compare the time to disease recurrence between participants who received LND vs participants who did not receive LND.
Use of adjuvant therapies | 2 years post-op
  T-test or the Wilcoxon rank-sum test will be applied to determine the rate of adjuvant therapies used between participants who received LND vs participants who did not receive LND.
Perioperative complications | 2 years post-op
  T-test or the Wilcoxon rank-sum test will be applied to determine the rate of perioperative complications between participants who received LND vs participants who did not receive LND.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Eltemamy, MD, Principal Investigator — Cleveland Clinic, Glickman Urological and Kidney Institute, Case Comprehensive Cancer Center; Adam Calaway, MD, MPH, Principal Investigator — University Hospitals Cleveland Medical Center, Urology Institute, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University of Florida Health Science Center, Gainesville, Florida
  - Southern Illinois University, Springfield, Illinois
  - University Hospitals Cleveland Medical Center, Urology Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Glickman Urological and Kidney Institute, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
This will be shared via a redcap database. All of the variables listed in the PRMC protocol and IRB application will be shared.
Time Frame: From when the trial starts (receives IRB approval and recruitment is initiated) until 1 year after the final participant finishes 2 year follow-up.
Access Criteria: This will be shared with the following people at UH PI, research coordinator, residents/fellows/other attendings who are included on the IRB at UH.